CLINICAL TRIAL: NCT06875427
Title: Comparing Preoperative Adductor Canal vs. No Block for Quality of Recovery After Anterior Cruciate Ligament Reconstruction in Patients Younger Than 18 Years of Age: A Randomized Controlled Feasibility Trial
Brief Title: ACB vs no Block for Pediatric ACL Reconstruction
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Isabella Jaramillo (Other)
Collaborators: McMaster University (Other)
Responsible Party: Sponsor-Investigator, Isabella Jaramillo, Principal Investigator, McMaster University
Organization: McMaster University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ssACB2024
Record Dates: First submitted 2024-11-27; First posted 2025-03-13 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Anterior Cruciate Ligament; Anterior Cruciate Ligament (ACL) Tear
Keywords: single-shot adductor canal block; anterior cruciate ligament reconstruction
MeSH Terms: conditions — Lacerations | interventions — Ropivacaine; Dexmedetomidine

STUDY DESIGN:
Intervention Model Description: Prospective randomized controlled feasibility study
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Research assistants involved in patient recruitment and follow-up.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Single-shot adductor canal block (Experimental): All the patients will receive a standardized general anesthetic technique, and adductor canal nerve block will be performed after induction using ropivacaine 2-2.5 mg/kg + dexmedetomidine 1 mcg/kg. IV placement in case of inhalational induction and airway secured.
  Interventions: Drug: Ropivacaine 2-2.5mg/kg + dexmedetomidine 1 mcg/kg delivered via a single-shot adductor canal block under ultrasound guidance
- Non-block (No Intervention): A general anesthetic will be performed as for the block group. NO nerve block will be performed. Dressing will be placed in the intended area of a block to maintain patient blinding.

INTERVENTIONS:
Drug: Ropivacaine 2-2.5mg/kg + dexmedetomidine 1 mcg/kg delivered via a single-shot adductor canal block under ultrasound guidance — The local anesthetic (ropivacaine) + dexmedetomidine will be administered via single-shot adductor canal block under ultrasound guidance
  Arms: Single-shot adductor canal block

SUMMARY:
The goal of this randomized controlled feasibility clinical trial is to assess the feasibility of conducting a randomized trial of adding a perioperative single-shot adductor canal block to standard of care general anesthesia compared to non-regional techniques in pediatric patients undergoing arthroscopic anterior cruciate ligament (ACL) reconstruction. The main clinical question it aims to answer is does ACB result in improved Quality of Recovery-15 questionnaire scores on postoperative day 2 , postoperative day 14, and postoperative day 42. Secondary questions this study will address are will use of a single-shot adductor canal block result in: less total opioid consumption; shorter post anesthetic care unit (PACU) length of stay; better pain scores at rest and with movement at time of postoperative phone call; and patient satisfaction score at 2 weeks (postoperative day 14). Researchers will compare the scores to patients undergoing the same surgery who will not have a single-shot ACB. All patients will receive the same pre-, peri-, and postoperative care with the exception of being randomized to block or no block. Participants will be asked to answer the Quality of Recovery-15 questionnaire and rate their pain on a scale of 0-10 on the day of surgery, at postoperative day 2 (by telephone) and at postoperative day 14 and postoperative day 42 during regular orthopedic clinic follow-up. Patients and caregivers will rate their satisfaction at postoperative day 42, using a 5-item Likert scale (ranging from completely dissatisfied to completely satisfied).

DETAILED DESCRIPTION:
Anterior cruciate ligament (ACL) injuries are becoming increasingly common among children and adolescents as they are engaging in contact sports at younger ages, which may contribute to a higher incidence of musculoskeletal injuries. This heightened susceptibility could be attributed to increased joint flexibility and potential immaturity in musculoskeletal development, with ACL reconstruction (ACLR) being the primary treatment approach. Effective pain management in the early postoperative phase is crucial, as it significantly impacts the ability to start rehabilitation and return to sports activities. Despite approximately 200,000 adolescents undergoing ACLR annually, there are no established benchmarks for pain management in this population, and significant variability exists in pain management practices in pediatric ACL reconstruction. Regional nerve blocks, such as femoral nerve blocks (FNBs), adductor canal blocks (ACBs), and sciatic nerve blocks (SNBs) are integral components of multimodal analgesia.

Recent research in the adult population has shown that multimodal analgesic strategies in arthroscopic surgeries can significantly reduce postoperative opioid consumption and improve quality of recovery.

In 2000, following the creation and initial clinical use of a 9-item Quality of Recovery (QoR) score, some authors introduced the 40-item QoR-40 and the shorter QoR-15. The QoR-15 scale provides a comprehensive assessment of postoperative recovery, with scores ranging from 0 (very poor QoR) to 150 (excellent QoR). Since then, the QoR-15 has emerged as the most commonly reported measure of patient-assessed quality of recovery after surgery, validated in the adult population.

The investigators plan to perform a prospective randomized controlled feasibility study comparing preoperative single-shot ACB to non-block in pediatric patients undergoing ambulatory arthroscopic ACL reconstruction. The investigators hypothesize that patients who received ACB preoperatively would have improved analgesia, fewer opioid-related adverse effects, greater patient satisfaction, and shorter PACU recovery times. Feasibility will be determined by enrollment rate, defined as the proportion of participants enrolled over the number of participants approached. We will declare feasibility if the enrollment rate is ≥ 80%.The primary clinical outcome variable is improvement in QoR-15 scores on POD2, POD14 and POD42.

ELIGIBILITY:
Inclusion Criteria:

* Patients ASA I, II and III
* 10-18 years of age
* scheduled for ACL reconstruction
* agreeable to regional block and follow-ups

Exclusion Criteria:

* Contraindications to adductor canal block.
* Patients with coagulopathies, preexisting neurologic deficit
* Significant comorbidities that may impact recovery or interfere with the study.
* Refusal to regional techniques.
* Moderate to severe cognitive deficit (patients who are unable to complete the questionnaire)
* Patients with history of malignant hyperthermia

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 38 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Change in Quality of Recovery scores | From day of surgery until end of study (postoperative day 42), collected at 4 timepoints: Day of surgery, postoperative day 2, postoperative day 14, postoperative day 42
  Assessed using the Quality of Recovery-15 (QoR-15) questionnaire, a validated 15-item questionnaire (patient survey). This questionnaire has 15 questions, each of which is answered on an 11-point Likert scale, where 10 = none of the time and 0 = All of the time. Final scores can range from 0 to 150. Scores will be compared between arms to see whether there is a difference in quality of recovery,
Enrollment rate | Period of recruitment is expected to be 12 months
  To determine feasibility, as defined as the proportion of participants enrolled over the number of participants approached. The investigators will declare feasibility if the enrollment rate is ≥ 80%.

SECONDARY OUTCOMES:
Pain control | From day of surgery until end of study (postoperative day 42), collected on postoperative day 0, postoperative day 2, postoperative day14 and postoperative day 42
  Patient will report pain on an 11-item numerical rating scale, where 0 = no pain and 10 = worst pain imaginable
Duration of post-anesthetic care unit stay | From time of time of hand-off to post-anesthetic care unit staff to discharge from the post-anesthetic care unit (usually by 2 hours [120 minutes])
  Duration of stay in post-anesthetic care unit, in minutes
Total opioid consumption | Day of surgery to postoperative day 14. Includes opioids used intraoperatively, in post-anesthetic care unit, and post-discharge.
  Milligrams of opioid per day, quantified as morphine equivalents. Data collected from electronic medical record and on patient visit at postoperative day 14 to clarify amount taken post-discharge.
Patient Satisfaction | From day of surgery to postoperative day 42. Patient is asked to rate satisfaction on day of surgery and again on postoperative day 42
  Patient asked to rate satisfaction regarding pain management on a 5-item scale, ranging from Very dissatisfied to Very satisfied
Caregiver Satisfaction | From day of surgery to postoperative day 42. Caregiver is asked to rate satisfaction on day of surgery and again on postoperative day 42
  Caregiver is asked to rate satisfaction regarding pain management on a 5-item scale, ranging from Very dissatisfied to Very satisfied
Hospital admission for any reason | Day of surgery until postoperative day 42
  Hospital admission for any reason (yes/no) will be recorded from electronic medical record and from interview with patient

CONTACTS AND LOCATIONS:
Locations (1):
- McMaster Children's Hospital, Hamilton Health Sciences, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data will be provided by PI on reasonable request once the data have been analyzed and published in a peer-reviewed journal
Supporting Information: Study Protocol
Time Frame: The investigators plan to publish the protocol in a peer-reviewed journal
Access Criteria: The IPD may be requested from the PI.